CLINICAL TRIAL: NCT04345094
Title: Randomized, Double-Blind Evaluation of Hexyresorcinol vs Hydroquinone for Photoaging
Brief Title: Evaluation of Hexyresorcinol vs Hydroquinone for Photoaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sytheon Ltd. (Industry)
Responsible Party: Principal Investigator, Ratan K. Chaudhuri, President, Sytheon Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HHSOL-1495-125
Record Dates: First submitted 2020-03-26; First posted 2020-04-14 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Photoaging
MeSH Terms: interventions — hydroquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator (Experimental): Emulsion containing 1% Hexylresourcinol
  Interventions: Other: Hexylresourcinol
- Intervention (Active Comparator): Emulsion containing 2% Hydroquinone
  Interventions: Other: Hydroquinone

INTERVENTIONS:
Other: Hexylresourcinol — Emulsion containing hexylresorcinol as an active
  Arms: Comparator
Other: Hydroquinone — Emulsions containing hydroquinone as an active
  Arms: Intervention

SUMMARY:
Photoaging is a common concern within the cosmeceutical industry with many products that are available. One frequently used product is hydroquinone that is used to even skin tone. However, hydroquinone has several shortcomings. The ingredient is controversial for its potential safety issues and it has been banned in Europe. An alternative ingredient that has emerged for its potential use is hexyresorcinol for evening skin tone. Additionally, hexylresorcinol may have other photoaging benefits such as the reduction in the appearance of fine lines.

Therefore, the aim of this study is to assess how hexyresorcinol may compare to the use of hydroquinone in the setting of photoaging.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 35-65 (limiting to females so that there is not heterogeneity with the influence of hormones. Also, females are a much larger user base of skin care products)
* Individuals who have not participated in any other clinical studies using the same test sites (face) and hand in the past 14 days
* Individuals with Fitzpatrick skin type I-IV
* No known medical conditions that, in the investigator's opinion, may interfere with study participation.

Exclusion Criteria:

* • Individuals who have been on any medication that has caused a change in skin pigmentation based on the opinion of the investigator

  * Individuals who have history of acute or chronic disease that would likely interfere with or increase the risk on study participation at the discretion of the investigator
  * Female volunteers who are pregnant or are actively breastfeeding or planning a pregnancy within two months. (There is no concern for risk to fetus but pregnancy can alter skin pigmentation)
  * Female volunteers who have started a new hormonal birth control agent or switched to a hormonal birth control agent within the past 60 days
  * Individuals who have had any medical or cosmetic procedure, such as laser resurfacing, or plastic surgery to the test site (face) within the last 6 months. This includes botulinum toxin, dermal fillers, collagen or other similar cosmetic procedure
  * Individuals who are currently using or during the past 30 days have used hydroquinone, or a retinoid such as Retin A, or other Rx/OTC Retinyl A.
  * Individuals who have used salicyclic acid, beta hydroxy acid, vitamins A, C, E in the 14 days prior to first visit.
  * Individuals with a known history of hypersensitivity to any ingredients to the cosmetic agent that is being assessed
  * Individuals who are pregnant, breast feeding or planning a pregnancy.
  * Individuals who have history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study at the discretion of the investigator

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
To assess the use of topical hexylresorcinol versus hydroquinone skin regimen on the objective appearance of skin photoaging - specifically appearance of pigment. | 12 weeks
  Assessed Through Skin Colorimeter (Validated Measurement Tool) - by melanin measurement on cheeks, hands, and face.
To assess the use of topical hexylresorcinol versus hydroquinone skin regimen on the clinical grading of appearance of skin photoaging - specifically appearance of pigment. | 12 weeks
  Pigment was assessed through clinical grading of 0 (none) to 3 (severe) scale by board-certified dermatologist of each side of the face.

SECONDARY OUTCOMES:
Observe and assess changes in the appearance of skin redness | 12 weeks
  Assessed using skin colorimeter (validated measurement tool) - by erythema measurement

OTHER OUTCOMES:
Subjective Tolerability Assessment | Assessed at Week 4, 8, and 12
  Assessed through subjective questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD, Principal Investigator — Pacific Skin Institute
Locations (1):
- Integrative skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will be published in a scientific journal with raw data made available to researchers upon request.

REFERENCES:
- [Derived] Wu H, Gabriel TA, Burney WA, Chambers CJ, Pan A, Sivamani RK. Prospective, randomized, double-blind clinical study of split-body comparison of topical hydroquinone and hexylresorcinol for skin pigment appearance. Arch Dermatol Res. 2023 Jul;315(5):1207-1214. doi: 10.1007/s00403-022-02514-0. Epub 2022 Dec 11. PMID 36502500